CLINICAL TRIAL: NCT04571892
Title: An Open-label, Single-arm, Single-dose Escalation and Multiple-dose Expansion Clinical Study of Cell Therapy to Evaluate the Tolerance, the Pharmacokinetic Characteristics, the Safety, and the Efficacy of ScTIL210 in the Treatment of Malignant Solid Tumors
Brief Title: A Clinical Study to Observe the Safety and Efficacy of ScTIL210 in the Treatment of Malignant Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ScTIL210-003-2020
Record Dates: First submitted 2020-08-18; First posted 2020-10-01 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Malignant Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ScTIL210 (Experimental): This trial is designed single arm. All the subjects enrolled will receive the experimental intervention, ScTIL210(Super circulating tumor infiltrating lymphocytes).
  Interventions: Biological: Super circulating tumor infiltrating lymphocytes(ScTIL)

INTERVENTIONS:
Biological: Super circulating tumor infiltrating lymphocytes(ScTIL) — Peripheral blood mononuclear cells (PBMCs) are used for cell preparation. PD-1(programmed death 1) positive T cells are isolated from peripheral blood by blood cell apheresis method and transduced with lentivirus loaded with "enhanced receptor" and "superamplification factor". The obtained ScTIL is used for one-time intravenous infusion.

SUMMARY:
An open-label, single-arm, single-dose escalation and multiple-dose expansion clinical study of cell therapy to observe and to evaluate the tolerance, the pharmacokinetic characteristics, the safety, and the efficacy of ScTIL210 in the treatment of malignant

ELIGIBILITY:
Inclusion Criteria:

* When patients meet ALL of the following requirements, they will be eligible to be recruited, at their own wills, to participate in the clinical study.

  1. Age ≥ 18 years old and ≤ 75 years old, regardless of gender;
  2. An expected survival duration of longer than 3 months;
  3. Patients with malignant solid tumor as confirmed by histology or cytology who failed in their prior standard therapies , or there is no recommended standard treatment, or a standard treatment is not applicable at this time;
  4. The proportion of PD-1 positive T lymphocytes to the total T lymphocytes is ≥ 18%. For patients who received PD-1 monoclonal antibody treatment within 4 weeks before screening, the proportion of PD-1 positive T to the total T lymphocytes is ≥ 12%;
  5. In accordance to RECIST version 1.1, there is at least one evaluable tumor focus for dose escalation phase; or there is at least one measurable tumor focus for dose expansion stage;
  6. ECOG physical status score of between 0 to 1;
  7. Sufficient bone marrow and organ function; Blood system:no transfusion or hematopoietic stimulating factor treatment within 14 days; Neutrophil count (ANC): ≥ 1.5 × 109/L; Platelet (PLT): ≥ 75 × 109/L; Hemoglobin (HB): ≥ 90 g/L; Absolute lymphocyte count (lym): ≥60% of the lower limit of normal range; Lymphocyte subsets:Percentage of B lymphocyte (CD19+) to the total lymphocyte of ≥9%； Liver function Total bilirubin (TBIL) : ≤ 1.5 × ULN Alanine aminotransferase (ALT): ≤ 3 × ULN; for patients with liver metastasis or liver cancer: ≤ 5 × ULN Aspartate aminotransferase (AST)： ≤ 3 × ULN; for patients with liver metastasis or liver cancer: ≤ 5 × ULN Renal function：Creatinine ≤ 1.5 × ULN Coagulation function：Activated partial thromboplastin time (APTT) ≤ 1.5 × ULN ；International normalized ratio (INR) ≤ 1.5 × ULN
  8. Eligible fertile patients (male and female) must agree to use reliable contraceptive methods (hormonal or barrier method or abstinence, etc.) with their partners during the trial and at least 90 days after the last medication; women of childbearing age (as defined in Appendix 8) must have a negative blood or urine pregnancy test within 7 days before the first use of the study drug;
  9. The subjects should be informed of the study before the trial and sign the written informed consent voluntarily.

Exclusion Criteria:

* When a patient has one of the following conditions, he or she will not be eligible to be recruited to the clinical study.

  1. Received chemotherapy, radiotherapy, biological therapy, endocrine therapy, immunotherapy, traditional chinese medicine with anti-tumor indications and other anti-tumor treatments within 2 weeks before apheresis procedure, except for the following items:

     1. Nitrosourea or mitomycin C treatment was within 6 weeks before apheresis;
     2. Oral administration of fluorouracil and small molecule targeted drugs was one week before apheresis.
  2. Received other unlisted clinical research drugs or treatments within 4 weeks before ;
  3. Major organ surgery (excluding puncture biopsy) or significant trauma occurred within 4 weeks before apheresis, or a surgery was scheduled during the trial period;
  4. Received systemic corticosteroids (prednisone > 10mg/day or equivalent dose of the similar drugs) or other immunosuppressants within 14 days before apheresis; Except for the following: topical, ocular, intra articular, nasal and inhaled glucocorticoids; short-term use of glucocorticoids for preventive treatment (e.g., prevention of contrast media allergy);
  5. Received immunomodulatory drugs, including but not limited to thymosin, interleukin-2, interferon, etc. within 14 days apheresis;
  6. Received live attenuated vaccine within 4 weeks before apheresis;
  7. The adverse reactions from previous anti-tumor therapy have not yet restored to CTCAE 5.0 grade evaluation of ≤1 (except for the toxicity without safety risk as judged by researchers such as alopecia).
  8. Central nervous system metastasis or meningeal metastasis with clinical symptoms, or other evidence indicating that the central nervous system metastasis or meningeal metastasis has not been controlled, as judged by researcher inappropriate to be recruited to the study;
  9. Patients with active infection within one week before apheresis and a systemic anti-infection treatment is essential at this time;
  10. History of immunodeficiency, including positive HIV antibody test;
  11. Hepatitis B (HBsAg positive and/or a positive hepatitis C antibody and/or a positive treponema pallidum antibody;
  12. Patients with progressive interstitial pneumonitis;
  13. Have a history of serious cardiovascular and cerebrovascular diseases, including but not limited to:

      1. There are serious cardiac arrhythmia or conduction abnormalities, such as 2-3 degree ventricular arrhythmia, , atrioventricular block, and so on.
      2. Acute coronary syndrome, congestive heart failure, aortic dissection, stroke or other cardiovascular and cerebrovascular events of grade 3 or above occurred within 6 months before the first administration.
      3. New York Heart Association (NYHA) defined cardiac function grade ≥ II or left ventricular ejection fraction (LVEF) of less than 50%, or as judged by other researchers to have a high risk of structural heart disease;
      4. Clinically uncontrollable hypertension.
  14. Patients with active or previous autoimmune diseases (such as systemic lupus erythematosus, rheumatoid arthritis, vasculitis, etc.) with active or previous autoimmune diseases (such as systemic lupus erythematosus, rheumatoid arthritis, vasculitis, etc.), excluding patients with clinically stable autoimmune thyroid disease and well controlled type I diabetes mellitus;
  15. Received immunotherapy and had Irae of grade 3 or above;
  16. The serous cavity exudation which could not be controlled clinically was not suitable for the study;
  17. Known alcohol or drug dependence;
  18. Mental disorder or poor compliance;
  19. Pregnant or lactating women;
  20. The researchers considered that the subjects were not suitable for the clinical study because of other serious systemic diseases or other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2020-10-15 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The safety of ScTIL210 | 24 weeks post infusion
  To assess if the ScTIL210 product will be safe to the subjects, as assessed by the incidence of treatment-related adverse events, in the treatment of malignant solid tumors.

SECONDARY OUTCOMES:
The in vivo dynamic variation of reinfused ScTIL210 | 24 weeks post infusion
  To assess the percentage of PD1 positive cell in total lymphocytes of peripheral blood along a series of time points after reinfusion of ScTIL210 as measured by flow cytometry.
The efficacy of ScTIL210 in the treatment of malignant solid tumors | 24 weeks post infusion
  To assess the clinical efficacy of ScTIL210 in the treatment of malignant solid tumors, as assessed by duration of response(DOR), i.e., time from complete remission (CR) or partial remission (PR) to disease progression (PD), or to death, or to last tumor evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, Ph.D., Principal Investigator — Shanghai Oriental Hospital
Locations (2):
- China (2):
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Shanghai Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality